CLINICAL TRIAL: NCT04692558
Title: Efficacy of Hyaluronic Acid on Connective Tissue Graft With Coronally Advanced Flap in the Treatment of Isolated Gingival Recession - A Randomized Controlled Clinical Trial.
Brief Title: Effect of Hyaluronic Acid on Gingival Recession Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 02_D012_102617
Record Dates: First submitted 2019-12-13; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HYALURONIC ACID (Experimental): CAF+CTG+HA
  Interventions: Biological: HYALURONIC ACID; Procedure: coronally advanved flap with connective tissue harvesting
- WITHOUT HYALURONIC ACID (Active Comparator): CAF+CTG
  Interventions: Procedure: coronally advanved flap with connective tissue harvesting

INTERVENTIONS:
Biological: HYALURONIC ACID — Hyaluronic acid will be applied on denuded root surface after reflection of isolated gingival recession.
  Other Names: HA
  Arms: HYALURONIC ACID
Procedure: coronally advanved flap with connective tissue harvesting — Coronally advanced flap surgery with connective tissue harvesting from palate
  Other Names: CAF+CTG

SUMMARY:
Gingival marginal tissue recession is the displacement of the soft tissue margin apical to the cementoenamel junction (CEJ) with exposure of the root surface. It is a common clinical finding in patients with high standards of oral hygiene and can be found in more than 90% of patients. Buccal exposure of roots leading to esthetic concerns and dentinal hypersensitivity are the most frequent reasons for patients to seek treatment for the same.

Gingival recession therapy is still challenging for clinicians. The ultimate goal of root coverage procedures is the complete coverage of the recession defect with an esthetic appearance comparable to adjacent healthy soft tissues in combination with physiological probing pocket depths.

Various treatment modalities have been put forth for the correction of gingival recession. These include free gingival autograft, subepithelial connective tissue graft (SCTG), coronally advanced flap (CAF) and various combinations. Coronally advanced flap (CAF) in conjunction with the connective tissue graft (CTG) is considered the gold standard of treatment of gingival recession due to its high predictability of the treatment results.

Several authors have explored the use of biological agents or like enamel matrix derivative (EMD), platelet-derived growth factor-BB (PDGF), fibroblast growth factor-2 (FGF-2), which are a group of proteins capable of inducing gene or cell activation for cell recruitment, matrix biosynthesis, and cellular differentiation, in an attempt to regenerate the lost periodontium to enhance its long term stability Hyaluronic acid (HA) is one such biologic agent that demonstrates future for periodontal regeneration. It is a major component of the extracellular matrix in almost all tissues. The primary role of HA is to bind water and to allow the transportation of key metabolites and therefore to maintain the structural and homeostatic integrity of these tissues. HA suppresses tissue breakdown activating metalloproteinase inhibitors. It represents one of the most hygroscopic molecules known in nature. As a physical background material, it functions as space filler, lubricant and a protein excluder as well. In vitro studies and animal studies have demonstrated that HA significantly increases the tensile strength of granulation tissue, stimulates clot formation, induces angiogenesis, increases osteogenesis, and does not interfere in the calcification nodules during bone formation. Furthermore, HA facilitates cell migration and differentiation during tissue formation and repair of both soft and hard tissues. It improves ligament cell viability and early osteogenic differentiation.

Considering the fact that HA has positive effects on wound healing, we hypothesized that it may also improve the results of root coverage by CAF+CTG. Therefore, the aim of this randomized controlled clinical trial (RCT) will be to evaluate the potential benefit of the adjunctive use of HA in combination with CAF+CTG and to compare the outcomes with CAF+CTG alone, when treating single Miller class I and class II/RT1gingival recessions.

DETAILED DESCRIPTION:
* After administration of local anesthesia
* Two oblique and divergent releasing incisions extending beyond the mucogingival junction (MGJ) will be performed. An intra-sulcular incision was performed at the buccal aspect of the involved tooth
* A second surgical site will be prepared to obtain the subepithelial CTG using single incision technique as described by Hurzeler and Weng.
* For the control group, only CAF+CTG will be performed. For the test group, cross-linked HA will be applied over the exposed root surface before the placement of CTG and CAF closure. HA will be presented as individual cartridge for single use only. For the application on the denuded root surface, the cartridge will be inserted into a cartridge syringe with 23G needles, as the fabricant recommended. HA will be applied on the root surface until completely covered, the harvested CTG will be placed and stabilized with sutures . Finally, the flap will be coronally displaced and sutured covering the CEJ. Interrupted sutures will be placed at the vertical releasing incisions in apical-coronal direction to reduce the tension and to facilitate the coronal displacement to perform the last coronal sling suture.
* Post-operative pain and edema will be controlled with anti-inflammatory drugs. Patients received Ibuprofen 400 mg thrice daily for 3 days19 and Amoxicillin 500mg thrice daily for 5 days.28 For patients allergic to penicillin Clindamycin 300 mg 4 times daily for 5 days will be prescribed.29
* A 60s rinse with 0.2% chlorhexidine gluconate was prescribed two times per day for the first 2 weeks.
* All participants will be instructed to intermittently apply an ice bag on the operated area.
* Participants will be recalled after a period of 14 days for suture removal. After this period patients will be reinstructed in mechanical cleaning of the treated teeth and use of a soft toothbrush and roll technique of brushing for one month.3
* Participants will be recalled for reinforcement of oral hygiene instructions and light debridement supragingivally will be carried out. Clinical parameters will be recorded at 6 weeks, 3 months and 6 months after surgical procedure.18

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to participate in the study.
* Age ≥ 18 to 55 years of age.
* Patients with healthy or treated periodontal condition.
* Full-mouth plaque score (FMPS) < 15%.
* Presence of at least one buccal recession (depth ≥ 2 mm) with no loss of interproximal attachment classified as Miller class I,II RT/1 in the anterior maxillary or mandibular area (central and lateral incisors, canine, and first and second premolars).
* Associated with esthetic problems and/or dental hypersensitivity.
* Gingival recession with at least 1 mm of keratinized tissue (KT) apical to the recession and thick gingival biotype (>0.8mm gingival thickness)

Exclusion Criteria:

* Active periodontal disease at sites (probing pocket depth < 4 mm and no bleeding on probing).
* Pregnant or lactating females.
* Tobacco smoking.
* Uncontrolled medical conditions.
* Untreated periodontal conditions.
* Use of systemic antibiotics in the past 3 months.
* Patients treated with any medication known to cause gingival hyperplasia.
* Drug and alcohol abuse.
* Occlusal interferences.
* History of mucogingival or periodontal surgery at the experimental site.
* Patients with a known hypersensitivity or allergy to hyaluronic acid.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
The difference in recession depth (RD) | 6 MOonths
  - measured as the distance from CEJ to the gingival margin.
complete root coverage (CRC) | 6 Months
  PERCENTAGE OF 100% ROOT COVERAGE
mean root coverage (MRC) | 6 Months
  MEASUREMENT OF AMOUNT OF COVERAGE OBTAINED OVER ALL
• Gingival recession width (GRW) | 6 Months
  measured as the distance between the mesial gingival margin (measurement will be recorded on a horizontal line tangential to the cementoenamel junction)
gingival thickness | 6 Months
  In the direct method, the tissue thickness is measured using a periodontal probe.
root coverage esthetic scores (RES). | 6 Months
  Root coverage esthetic score: a system to evaluate the esthetic outcome of the treatment of gingival recession through evaluation of clinical cases. ... This score evaluates five variables: level of the gingival margin, marginal tissue contour, soft tissue texture, mucogingival junction alignment, and gingival color.

SECONDARY OUTCOMES:
Pocket probing depth | 6 Months
  Measure the pocket depth of the groove between your gums and teeth by placing a dental probe beside your tooth beneath your gumline, usually at several sites throughout your mouth. In a healthy mouth, the pocket depth is usually between 1 and 3 millimeters (mm). Pockets deeper than 4 mm may indicate periodontitis.
clinical attachment level (CAL) | 6 Months
  CAL is calculated from a fixed reference point (cementoenamel junction or CEJ), and it is computed by calculating the distance from the CEJ to the base of the pocket. When the gingival margin is coronal to the CEJ, you subtract (from the probing depth) the distance from the CEJ to the gingival margin.
width of keratinized tissue (KTW) | 6 Months
  Place your probe on the outside of the tissue and measure from the gingival margin to the mucogingival junction. Now measure the sulcus or pocket depth (probing depth). Subtract the probing depth from the outside measurement of the gingiva, and you will have the width of attached gingiva.
plaque index (PI) | 6 Months
  Plaque Index = (2+1+1+2) / 4 = 1.5, according to the plaque index system this means the plaque index for the tooth is moderate accumulation of soft deposit within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye.
gingival index (GI) | 6 Months
  The Gingival Index (Löe and Silness, 1963) was created for the assessment of the gingival condition and records qualitative changes in the gingiva. It scores the marginal and interproximal tissues separately on the basis of 0 to 3.
bleeding index (BI) | 6 Months
  The gingival bleeding index of Ainamo J and Bay I was developed as an easy and suitable way for assessing a patient's progress in Plaque control. The presence or absence of gingival bleeding is determined by gentle probing of the gingival crevice with a periodontal probe. The appearance of bleeding within 10 seconds indicates a positive score, which is expressed as percentage of the total number of gingival margin examined.
VAS scale for pain and esthetic | 14 days
  Esthetics-post treatment outcomes. 0-Not Satisfied 10- Very Satisfied
The Wound healing index | 14 days
  Wound Healing Index (Huang et al 2005) Score 1 Uneventful healing with no gingival edema, erythema, suppuration, patient discomfort or flap dehiscence.
  Score 2 Uneventful healing with slight gingival edema, erythema, patient discomfort, or flap dehiscence, but no suppuration.
  Score 3 Poor wound healing with significant gingival edema, erythema, patient discomfort, flap dehiscence, or any suppuration.

CONTACTS AND LOCATIONS:
Overall Officials: PRABHUJI MLV, MDS, Study Director — Krishnadevaraya College of Dental Sciences & Hospital
Locations (1):
- Krishnadevaray College of Dental Science and Hospital, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pilloni A, Schmidlin PR, Sahrmann P, Sculean A, Rojas MA. Effectiveness of adjunctive hyaluronic acid application in coronally advanced flap in Miller class I single gingival recession sites: a randomized controlled clinical trial. Clin Oral Investig. 2019 Mar;23(3):1133-1141. doi: 10.1007/s00784-018-2537-4. Epub 2018 Jun 30. PMID 29961138
- [Background] Kumar R, Srinivas M, Pai J, Suragimath G, Prasad K, Polepalle T. Efficacy of hyaluronic acid (hyaluronan) in root coverage procedures as an adjunct to coronally advanced flap in Millers Class I recession: A clinical study. J Indian Soc Periodontol. 2014 Nov-Dec;18(6):746-50. doi: 10.4103/0972-124X.147411. PMID 25624632